CLINICAL TRIAL: NCT03696355
Title: Phase I Study of GDC-0084, a Brain-Penetrant PI3 Kinase/mTOR Inhibitor, in Pediatric Patients With Newly Diagnosed Diffuse Intrinsic Pontine Glioma or Diffuse Midline Gliomas After Radiation Therapy
Brief Title: Study of GDC-0084 in Pediatric Patients With Newly Diagnosed Diffuse Intrinsic Pontine Glioma or Diffuse Midline Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Kazia Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJPI3K; NCI-2018-02268 (Registry Identifier: NCI Clinical Trial Registration)
Record Dates: First submitted 2018-10-03; First posted 2018-10-04 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: Anaplastic Astrocytoma; Atypical Brainstem Glioma; Brain Cancer; Brain Stem Glioma; Brain Tumors in Children; Diffuse Intrinsic Pontine Glioma; Diffuse Midline Glioma; Glioblastoma; H3 K27M mutant; Newly Diagnosed; Non-brainstem Midline Glioma; Pediatric Brain Tumor; Radiation Therapy; St. Jude Brain Tumor Studies; St. Jude Studies; St. Jude Treatment
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Brain Neoplasms; Diffuse Intrinsic Pontine Glioma; Glioblastoma | interventions — GDC-0084; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stratum A1 (Experimental): Dose Escalation Phase:
  Four to 12 weeks after the completion of standard RT, subjects who are able to swallow capsules will receive single-agent oral GDC-0084 at one of the 4 dose levels once daily in cycles of 28 days. During cycle 1 only, a single dose of GDC-0084 will be withheld on day 2, for a total of 27 doses. Treatment may be continued for up to 24 months (26 cycles) in the absence of disease progression or unacceptable toxicity.
  Dose Expansion Phase
  Four to 12 weeks after the completion of standard RT, subjects who are able to swallow capsules will receive the MTD dose established in the Stratum A dose escalation phase. Subjects who completed the first course of therapy may take GDC-0084 as an open capsule sprinkled in purée such as applesauce. Treatment may be continued for up to 24 months (26 cycles) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: GDC-0084; Radiation: radiation therapy
- Stratum A2 (Experimental): Four to 12 weeks after the completion of standard RT, subjects will received the MTD dose established in the Stratum A1 dose escalation phase. Subjects who are unable to swallow capsules will initially be enrolled until the Stratum A1 expansion cohort is filled. Once the Stratum A1 expansion cohort has been filled, both subjects who are able to swallow capsules and those unable to swallow capsules may be enrolled. Subjects who are unable to swallow capsules will take GDC-0084 as an open capsule sprinkled in purée such as applesauce. Subjects who have completed the first course of therapy and are able to swallow capsules may take GDC-0084 as capsules. Treatment may be continued for up to 24 months (26 cycles) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: GDC-0084; Radiation: radiation therapy

INTERVENTIONS:
Drug: GDC-0084 — Given PO
Radiation: radiation therapy — Both photon and proton therapy modalities will be allowed.
  Other Names: irradiation; radiotherapy; radiation; external beam radiation therapy (EBRT)

SUMMARY:
Pediatric high-grade gliomas are highly aggressive and treatment options are limited. The purpose of this first-in-pediatrics study is to examine the safety, tolerability, and pharmacokinetics of GDC-0084 and to estimate its maximum tolerated dose (MTD) when administered to pediatric patients with diffuse intrinsic pontine glioma (DIPG) or other diffuse midline H3 K27M-mutant gliomas after they have received radiation therapy (RT). GDC-0084 is a brain-penetrant inhibitor of a growth-promoting cell signaling pathway that is dysregulated in the majority of diffuse midline glioma tumor cells. This study is also designed to enable a preliminary assessment of the antitumor activity of single-agent GDC-0084, in the hope of enabling rational combination therapy with systemic therapy and/or radiation therapy (RT) in this patient population, which is in desperate need of therapeutic advances.

Primary Objectives

1. To estimate the maximum tolerated dose (MTD) and/or the recommended phase 2 dosage (RP2D) of GDC-0084 in pediatric patients with newly diagnosed diffuse midline glioma, including diffuse intrinsic pontine glioma (DIPG)
2. To define and describe the toxicities associated with administering GDC-0084 after radiation therapy (RT) in a pediatric population
3. To characterize the pharmacokinetics of GDC-0084 in a pediatric population

Secondary Objectives

1. To estimate the rate and duration of radiographic response in patients with newly diagnosed DIPG or other diffuse midline glioma treated with RT followed by GDC-0084
2. To estimate the progression-free survival (PFS) and overall survival (OS) distributions for patients with newly diagnosed DIPG or other diffuse midline glioma treated with RT followed by GDC-0084

DETAILED DESCRIPTION:
There are two research strata: Stratum A1 and Stratum A2. All subjects will receive standard RT no later than 14 days after study enrollment and no later than 42 days after the date of radiographic diagnosis or surgery, whichever date is the later. Four to 12 weeks after the completion of standard RT, subjects without radiographic evidence of progression will receive single-agent oral GDC-0084 once daily in cycles of 28 days. Treatment may be continued for up to 2 years in the absence of disease progression or unacceptable toxicity.

Subjects enrolled on Stratum A1 will be enrolled on the dose-escalation phase of the study. Up to 4 different dose levels will be evaluated: Dose level 0, 21 mg/m2; Dose level 1, 27 mg/m2; Dose level 2, 35 mg/m2; and Dose level 3, 45 mg/m2. The Rolling 6 design will be used to determine the maximum tolerated dose (MTD)/recommended phase 2 dosage (RP2D) of GDC-0084.

Subjects enrolled on Stratum A1 must be able to swallow capsules during the first cycle of therapy (the dose-limiting toxicity (DLT) evaluation period). Subjects who complete the DLT evaluation period and are no longer able to swallow the whole capsule may take GDC-0084 opened, sprinkled in purée. Additionally, subjects who gain the ability to swallow whole capsules after initially receiving the opened formulation and have completed the DLT evaluation period may transition to the whole capsule formulation. Subjects who change administration methods after course 1 will have mandatory intrapatient pharmacokinetic studies performed. Subjects enrolled on Stratum A1 who are no longer able to swallow whole capsules of GDC-0084 during the DLT evaluation period (cycle 1) will be taken off treatment.

Once the MTD has been established in Stratum A1, the Stratum A1 expansion cohort and Stratum A2 will open simultaneously. Subjects enrolled on the Stratum A1 expansion cohort will be required to swallow capsules. Subjects enrolled on Stratum A2 will be restricted to subjects who are unable to swallow capsules until the Stratum A1 expansion cohort is filled. Once the Stratum A1 expansion cohort has been filled, both subjects who are able to swallow capsules and those unable to swallow capsules may be enrolled on Stratum A2. Subjects enrolled on Stratum A2 who are unable to swallow capsules will take GDC-0084 as an open capsule sprinkled in purée and will undergo mandatory interpatient pharmacokinetic studies.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 2 years and less than 22 years at the time of enrollment
* Subjects must have one of the following newly diagnosed tumors:

  * Non-biopsied typical DIPG, defined as a tumor with a pontine epicenter and diffuse intrinsic involvement of the pons. These subjects are eligible without histologic confirmation.
  * Biopsied typical DIPG: WHO grade II diffuse astrocytoma (IDH WT or IDH NOS), WHO grade III anaplastic astrocytoma (IDH WT or IDH NOS), WHO grade IV glioblastoma (IDH WT or IDH NOS), or diffuse midline glioma, H3 K27M mutant. Subjects with a typical DIPG who undergo a biopsy may be eligible for the study if the tumor does not harbor the H3 K27M mutation, yet eligibility is restricted to diffuse astrocytoma, anaplastic astrocytoma or glioblastoma, IDH WT or IDH NOS, tumors.
  * Atypical brainstem glioma: diffuse midline glioma, H3 K27M mutant.
  * Non-brainstem midline glioma, defined as tumors with an epicenter within midline structures, including the thalamus, spinal cord, and cerebellum: diffuse midline glioma, H3 K27M mutant.
* Subjects must have localized, non-metastatic disease; MRI of spine must be performed if disseminated disease is suspected by the treating physician.
* Subjects must be able to start radiation therapy no later than 42 days after radiographic diagnosis or surgery, whichever date is later.
* Performance score ≥ 50 (Lansky for research subjects aged 16 years or younger and Karnofsky for subjects older than 16 years). Subjects who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Subjects must not have received any prior therapy, including prior treatment with a PI3 kinase, mTOR, or PI3K/mTOR inhibitor, other than surgery and/or steroids.
* Subjects must have adequate organ function documented at the time of study enrollment as follows:

  * Bone marrow: Hemoglobin ≥ 8g/dL [may have received packed red blood cell transfusion], absolute neutrophil count (ANC) ≥ 1000/mm^3, platelets ≥ 50,000/mm^3 [transfusion independent].
  * Renal: Normal serum creatinine based on age (Age 2 to ≤5: 0.8; Age >5 to <10: 1.0; Age >10 to <15: 1.2; Age ≥15: 1.5) or GFR ≥ 70 mL/min/1.73m^2
  * Hepatic: ALT and AST < 3 × the institutional upper limit of normal (ULN), total bilirubin concentration < 1.5 x the institutional ULN, albumin ≥ 2g/dL.
* Shortening fraction of ≥ 27% by ECHO or ejection fraction of ≥ 50% by gated radionuclide study.
* Subjects must not have congenital long QT syndrome and QTc < 500 ms.
* Subjects must not require the use of any CYP34A-inducing or -inhibiting agents, with the exception of corticosteroids.
* Female subjects of childbearing potential must not be pregnant or breastfeeding a child. Female subjects of childbearing potential aged 10 years or older must have a negative serum or urine pregnancy test.
* Subjects of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control, which can be abstinence, while being treated on this study and for 3 additional months after completion of therapy.
* Informed consent: All subjects and/or their parents or legally authorized representatives must sign a written consent. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

* Subjects with evidence of tumor infiltration of three or more cerebral lobes on diagnostic MRI.
* Subjects with any clinically significant, unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic, or other organ dysfunction) that would compromise the subject's ability to tolerate protocol therapy or would probably interfere with the study procedures or results.
* Diabetic subjects who require insulin therapy.
* Subject with a history of clinically significant, uncontrolled heart disease and/or repolarization abnormalities as documented by a standard 12-lead ECG.
* Subjects receiving any other anticancer (glucocorticoids are acceptable) or investigational drug therapy.
* Subjects unable to return for follow-up visits or obtain follow-up studies required to assess toxicity of therapy.
* Subjects with disseminated disease.
* Pregnant subjects or subjects breast-feeding a child.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2022-09-04 (Actual)

PRIMARY OUTCOMES:
Estimate the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of GDC-0084 after standard-of-care radiation therapy (RT) | 1 month after start of GDC-0084 treatment
  The MTD is empirically defined as the highest dose level at which six patients have been treated with at most one patient experiencing a dose-limiting toxicity (DLT) and the next higher dose level has been determined to be too toxic. The MTD estimate will not be available if the lowest dose level studied is too toxic or the highest dose level studied is considered safe. In the latter case, the highest studied safe dose may be considered as the recommended phase 2 dose (RP2D). The MTD estimation will be limited to evaluable patients and toxicity assessments from course 1 (28 days).
Incidence of adverse events at least possibly associated with GDC-0084 after RT by stratum | Up to 2 years after start of GDC-0084 treatment
  Adverse event data will be summarized in tables by dose level.
Pharmacokinetics of GDC-0084 by stratum | GDC-0084 treatment course 1 days 1 and 28
  GDC-0084 area under the curve (AUC0-∞) is estimated based on course 1 day 1 (C1D1) PK samples, and AUC0-24 based on course 1 day 28 (C1D28) PK samples.

SECONDARY OUTCOMES:
Rate of best overall response by stratum | Up to 1 year after completion of GDC-0084 treatment
  The best overall response is the best response recorded between the start of GDC-0084 treatment and the earliest of initiation of alternative therapy or disease progression/recurrence. Best responses include complete response (CR), partial response (PR), and stable disease (SD). The best response is unknown if the patient does not qualify for a best response of progressive disease and if all objective statuses after the first determination and before progression are unknown.
Duration of best overall response by stratum | Up to 1 year after completion of GDC-0084 treatment
  The duration of best overall response is measured from the time the measurement criteria are met for CR, PR, or SD (whichever is recorded first) until the first day on which recurrent or progressive disease is objectively documented.
Progression-free survival for patients treated with GDC-0084 after RT | Up to 3 years from diagnosis
  Progression-free survival (PFS) is defined from the time of diagnosis until disease progression or until death from any cause for patients who experience an event and until the date of last follow-up for those who are alive and progression free at the time of analysis. PFS is estimated by Kaplan-Meier approach and median PFS is reported.
Overall survival for patients treated with GDC-0084 after RT | Up to 3 years from diagnosis
  Overall survival (OS) is defined from the time of diagnosis until death from any cause for patients who experience an event and until the date of last follow-up for those who are alive at the time of analysis. OS is estimated by Kaplan-Meier approach and median OS is reported.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Tinkle, MD, PhD, Principal Investigator — St. Jude Children's Research Hospital; Amar Gajjar, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols
- See also: St. Jude Brain Tumor Studies — http://www.stjude.org/research/clinical-trials.html#c671955e2f6ffa4a5f9cd8cf39931465e1f28ef99042a579a1474aa7f29de3b5=2